CLINICAL TRIAL: NCT03248830
Title: Evaluation of Non-invasive Hemoglobin Monitoring in Children With Congenital Heart Diseases
Brief Title: Non-invasive Hemoglobin Monitoring in Congenital Heart Diseased Children
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Other Study IDs: N-99-2017
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: radical-7 pulse co-oximeter — Radical-7 pulse co-oximter will be applied to the patient through a special probe attached the the patient digit to measure blood hemoglobin
  Other Names: Masimo pulse co-oximeter

SUMMARY:
The investigators will evaluate the accuracy of non-invasive hemoglobin monitor (Sp-Hb) compared to traditional laboratory hemoglobin (Lab-Hb) in children with congenital heart disease. The investigators will also compare the accuracy of Sp-Hb in cyanotic children to acyanotic children.

DETAILED DESCRIPTION:
Blood hemoglobin is measured daily in clinical practice. Laboratory measurement (Lab-Hb) of is the gold standard for assessment of blood hemoglobin. Recently, non-invasive monitors had been introduced. Non-invasive measurement of hemoglobin (Sp-Hb) would save time and minimize the risk of infection. Blood sampling in children is usually more difficult and stressful; moreover, it also carries the risk of iatrogenic anemia.

Radical-7 (Masimo corporation, Irvine, CA) is a device that operates using the principle of co-oximetry . Radical-7 had been validated in various clinical purposes. Measurement of blood hemoglobin is an important application for Radical-7 device. Non-invasive hemoglobin (Sp-Hb) measurement has been frequently validated in adults; as well as in pediatric patients; however, its accuracy in children with congenital heart disease was not investigated. Congenital heart disease infants usually undergo major operations and frequently need transfusion of blood. Moreover, these patients have special circulatory physiology that might impact the device accuracy. It had been recently reported that the performance of co-oximetry in congenital heart disease children is poor in measurement of oxygen saturation specially at oxygen saturation under 75%; however, its accuracy in measurement of hemoglobin was not investigated yet. In this study, the investigators will evaluate the accuracy of Sp-Hb compared to traditional Lab-Hb in children with congenital heart disease. the investigators will also compare the accuracy of Sp-Hb in cyanotic children to acyanotic children.

ELIGIBILITY:
Inclusion Criteria:

* infants and children less than 8 years
* with congenital heart disease

Exclusion Criteria:

* refusal of the patient surrogate to share in the study

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will include children less than 8 years with congenital hear diseases scheduled for surgery or endo-vascular iintervention
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
non-invasive hemoglobin | 5 hours
  the value of hemoglobin measured by radical-7 device in g/dL

SECONDARY OUTCOMES:
laboratory hemoglobin | 5 hours
  the value of hemoglobin measured from a blood sample in the laboratory in g/dL
perfusion index | 5 hours
  the percentage of perfusion index measured by radical-7 device
plethysmography variability index | 5 hours
  the percentage of plethysmography variability index measured by radical-7 device
systolic blood pressure | 5 hours
  systolic blood pressure measured in mmHg
diastolic blood pressure | 5 hours
  diastolic blood pressure measured in mmHg
oxygen saturation from radical-7 device | 5 hours
  oxygen saturation measured by radical-7 device
oxygen saturation from arterial blood gases | 5 hours
  oxygen saturation measured from arterial blood gases
heart rate | 5 hours
  number of heart beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No